CLINICAL TRIAL: NCT03865940
Title: A Randomized, Double-Blind, 2-Way Crossover Trial to Assess the Efficacy of Guanfacine and Lidocaine Combination Versus Lidocaine Alone in Trigeminal Nerve Block for Pain Management in Painful Trigeminal Neuropathy Patients
Brief Title: Efficacy of Guanfacine and Lidocaine Combination in Trigeminal Nerve Block for Pain Management in Trigeminal Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Tigran Keseyan, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TN
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Lidocaine; Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lidocaine then Lidocaine + Guanfacine (Experimental): Trigeminal nerve block will be performed with injection of 6 mL of 1% lidocaine (Day 1).
  Patient will return between Day 15-28 and trigeminal nerve block will be performed with injection of 6 mL of 1% lidocaine + 250 mcg guanfacine.
  Interventions: Drug: Lidocaine; Drug: Guanfacine
- Lidocaine + Guanfacine then Lidocaine (Experimental): Trigeminal nerve block will be performed with injection of 6 mL of 1% lidocaine + 250 mcg guanfacine (Day 1).
  Patient will return between Day 15-28 and trigeminal nerve block will be performed with injection of 6 mL of 1% lidocaine.
  Interventions: Drug: Lidocaine; Drug: Guanfacine

INTERVENTIONS:
Drug: Lidocaine — 6 mL of 1% lidocaine
  Other Names: Xylocaine
Drug: Guanfacine — 250 mcg

SUMMARY:
A phenome-wide association study (PheWAS) identified an association between a loss of function variant in the human alpha 2B adrenergic receptor gene and trigeminal nerve disorders. Guanfacine is the oldest alpha-2 adrenergic agonist in clinical use and is approved for hypertension and attention deficit hyperactivity disorder. We hypothesize that guanfacine will be an effective adjunct to lidocaine for the treatment of neuropathic pain by enhancing and prolonging pain relief due to its activation of alpha-2 adrenergic receptors. The objectives of the study will be to evaluate the efficacy and safety of guanfacine in combination with lidocaine for trigeminal nerve block procedures for pain management in trigeminal neuralgia patients. This study will evaluate the efficacy of guanfacine in reducing acute pain and extending duration of pain relief when delivered in combination with lidocaine as a trigeminal nerve block, measured by Visual Analog Scale (VAS) data collected at specific time points after each injection.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and read English
* History of painful trigeminal neuropathy with persistent background facial pain severity > 5/10 on VAS
* Experience pain with a score of greater than 5 on a 0-10 scale (VAS) in the previous 24 hours before procedural treatment and at the time of procedural treatment.
* Eligible for trigeminal nerve block procedure and have not had a trigeminal nerve block procedure for pain management prior to the enrollment in the current study.
* Able to provide informed consent.

Exclusion Criteria:

* Presence of a significant structural lesion (e.g., tumor) as the cause of pain as shown in at least one neuroimaging study.
* Current diagnosis of fibromyalgia, temporomandibular disorders (TMD), odontogenic pain or other orofacial pain deemed unrelated to the trigeminal nerve as the origin.
* Allergy or any other hypersensitivity reactions to guanfacine or lidocaine or local anesthetic of the amide type, or to both iodinated contrast and gadolinium contrast.
* Females who are pregnant or breastfeeding and/or plan to become pregnant or to breastfeed during study participation.
* Participation in another investigational drug study within 30 days before randomization.
* Inability to understand the requirements of the study, inability to abide by the study restrictions, inability to fill out the questionnaires, or inability to return for the required treatments.
* Any clinically significant medical or surgical condition that in the investigator's opinion could interfere with the administration of study drug, interpretation of study results, or compromise the safety or well-being of the subject (i.e. infection, unable to stop anticoagulants).
* No reliable access to telephone service to allow for contact with study personnel.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tigran Kesayan, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meier SE, Orr MB, Shotwell MS, Jerome RN, Shirey-Rice JK, Pulley JM, Edwards DA, Toye AD, Mishra P, Kesayan T. Enhanced pain relief with guanfacine as an adjuvant for trigeminal nerve blocks: insights from a PheWAS-guided randomized controlled study. Pain Med. 2025 Oct 1;26(10):643-654. doi: 10.1093/pm/pnaf054. PMID 40326696

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine Then Lidocaine + Guanfacine: Trigeminal nerve block will be performed with injection of 6 mL of 1% lidocaine (Day 1).
  Patient will return between Day 15-28 and trigeminal nerve block will be performed with injection of 6 mL of 1% lidocaine + 250 mcg guanfacine.
  Lidocaine: 6 mL of 1% lidocaine
  Guanfacine: 250 mcg
- Lidocaine + Guanfacine Then Lidocaine: Trigeminal nerve block will be performed with injection of 6 mL of 1% lidocaine + 250 mcg guanfacine (Day 1).
  Patient will return between Day 15-28 and trigeminal nerve block will be performed with injection of 6 mL of 1% lidocaine.
  Lidocaine: 6 mL of 1% lidocaine
  Guanfacine: 250 mcg
Period: First Intervention (14 Days)
Arm/Group | Lidocaine Then Lidocaine + Guanfacine | Lidocaine + Guanfacine Then Lidocaine
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0
Period: Washout Period (14 Days)
Arm/Group | Lidocaine Then Lidocaine + Guanfacine | Lidocaine + Guanfacine Then Lidocaine
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Lidocaine Then Lidocaine + Guanfacine | Lidocaine + Guanfacine Then Lidocaine
Started | 18 | 19
Completed | 10 | 18
Not Completed | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Then Lidocaine + Guanfacine | Lidocaine + Guanfacine Then Lidocaine | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.5 [47.1 to 64.6] | 60.1 [49.7 to 69.2] | 60.0 [47.8 to 68.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 19 | 35
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Time to Return to Baseline Pain After Injection.
Description: Time (hours) until pain returns to baseline number.
Time Frame: up to 2 weeks
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Lidocaine Alone: Data from injection where participants received an injection of lidocaine ALONE.
- Lidocaine + Guanfacine: Data from injection where participants received lidocaine + guanfacine.
Arm/Group | Lidocaine Alone | Lidocaine + Guanfacine
Number analyzed (Participants) | 36 | 28
hours | 8 [4 to 120] | 5 [5 to 168]
Statistical Analysis 1: Comparison: Lidocaine Alone vs Lidocaine + Guanfacine; Test type: Superiority; p = 0.374, Regression, Cox — P-values less than 0.05 considered significant; Testing null hypothesis that guanfacine has no effect on time from injection to return to baseline

2. Secondary Outcome: Pain Intensity in Follow-Up
Description: Pain Intensity after treatment measured throughout the 8-hour follow-up period on a visual analog scale (VAS) from 0 to 10, where 0 is the least pain and 10 is the most pain.
Time Frame: 8 hours
Population: The overall number of participants analyzed corresponds with how many participants were injected; however, not every participant responded at every timepoint. Therefore, only recorded responses at each timeline were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine Alone | Lidocaine + Guanfacine
Number analyzed (Participants) | 36 | 28
score on a scale
  0 hours | 6.75 (1.56) | 6.63 (1.43)
  0.5 hours: number analyzed (Participants) | 35 | 26
  0.5 hours | 1.91 (2.31) | 1.88 (2.72)
  1 hour: number analyzed (Participants) | 34 | 26
  1 hour | 2.24 (2.2) | 1.54 (2.25)
  1.5 hours: number analyzed (Participants) | 30 | 24
  1.5 hours | 2.83 (2.6) | 1.42 (1.98)
  2 hours: number analyzed (Participants) | 30 | 27
  2 hours | 2.47 (2.26) | 1.81 (2.11)
  2.5 hours: number analyzed (Participants) | 30 | 24
  2.5 hours | 2.7 (2.53) | 2.21 (2.45)
  3 hours: number analyzed (Participants) | 31 | 25
  3 hours | 2.84 (2.38) | 2.4 (2.61)
  3.5 hours: number analyzed (Participants) | 30 | 24
  3.5 hours | 3.03 (2.37) | 2.38 (2.45)
  4 hours: number analyzed (Participants) | 31 | 26
  4 hours | 2.74 (2.18) | 2.04 (2.49)
  4.5 hours: number analyzed (Participants) | 31 | 21
  4.5 hours | 2.79 (2.18) | 2.29 (2.41)
  5 hours: number analyzed (Participants) | 31 | 26
  5 hours | 3.65 (2.12) | 2.58 (2.44)
  5.5 hours: number analyzed (Participants) | 29 | 25
  5.5 hours | 3.69 (2.14) | 3.0 (2.81)
  6 hours: number analyzed (Participants) | 32 | 27
  6 hours | 3.31 (2.24) | 2.67 (2.45)
  6.5 hours: number analyzed (Participants) | 31 | 26
  6.5 hours | 3.42 (2.17) | 2.81 (2.23)
  7 hours: number analyzed (Participants) | 29 | 24
  7 hours | 3.76 (2.4) | 2.79 (2.17)
  7.5 hours: number analyzed (Participants) | 27 | 26
  7.5 hours | 3.52 (2.65) | 2.85 (2.19)
  8 hours | 3.56 (2.53) | 2.68 (2.25)
Statistical Analysis 1: Comparison: Lidocaine Alone vs Lidocaine + Guanfacine; Test type: Superiority; p < 0.001, Regression, Logistic — P-values less than 0.05 considered significant; Analysis adjusted for pre-injection score and accounted for repeated measures. Effect of study drug was tested using a four degree-of-freedom test

3. Secondary Outcome: Quality of Life, Physical Health
Description: Participant Quality of Life as measured by the PROMIS Global Health -10 SF during the 14-day follow-up. The scores reported are T-scores. The T-score rescales the raw sum score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean and a person with a T-score of 60 is one SD above the mean.
  For the Physical Health subscale, raw scores are converted into t-scores ranging from 16.2 to 67.7 and higher t-scores are indicative of better overall physical health.
Time Frame: 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lidocaine Alone | Lidocaine + Guanfacine
Number analyzed (Participants) | 36 | 28
T-score
  Day 0 | 40.35 (6.66) | 39.86 (6.07)
  Day 7: number analyzed (Participants) | 33 | 28
  Day 7 | 42.88 (6.47) | 43.2 (6.3)
  Day 14: number analyzed (Participants) | 31 | 28
  Day 14 | 42.83 (7.89) | 41.67 (7.16)
Statistical Analysis 1: Comparison: Lidocaine Alone vs Lidocaine + Guanfacine; Test type: Superiority; p = 0.775, Regression, Linear; The analysis adjusted for pre-injection score and accounted for repeat measures.The results of the analyses tested using a two degree-of-freedom test

4. Secondary Outcome: Quality of Life, Mental Health
Description: Participant Quality of Life as measured by the PROMIS Global Health -10 SF during the 14-day follow-up. The scores reported are T-scores. The T-score rescales the raw sum score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean and a person with a T-score of 60 is one SD above the mean.
  In this Mental Health subscale, raw scores are converted into t-scores ranging from 21.2 to 67.6, where higher t-scores are indicative of better overall physical health.
Time Frame: 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lidocaine Alone | Lidocaine + Guanfacine
Number analyzed (Participants) | 36 | 28
T-score
  Day 0 | 44.98 (10.47) | 44.4 (8.93)
  Day 7: number analyzed (Participants) | 33 | 27
  Day 7 | 44.34 (8.42) | 46.07 (8.42)
  Day 14: number analyzed (Participants) | 31 | 28
  Day 14 | 43.78 (7.91) | 45.72 (9.91)
Statistical Analysis 1: Comparison: Lidocaine Alone vs Lidocaine + Guanfacine; Test type: Superiority; p = 0.099, Regression, Linear; [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: Frequency of Nerve Pain Attacks
Description: Frequency of nerve pain attacks during the 14-day follow-up period. Pain frequency was recorded numerically as 0 - None (no pain), 1 - Weekly, 2 - Daily, 3 - Hourly, and 4 - Constant pain. Data was not collected at baseline, only at Day 7 and Day 14.
Time Frame: 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Alone | Lidocaine + Guanfacine
Number analyzed (Participants) | 36 | 28
units on a scale
  Day 7: number analyzed (Participants) | 33 | 27
  Day 7 | 3.64 (1.11) | 3.70 (1.17)
  Day 14: number analyzed (Participants) | 31 | 27
  Day 14 | 3.61 (1.15) | 3.81 (0.83)
Statistical Analysis 1: Comparison: Lidocaine Alone vs Lidocaine + Guanfacine; Test type: Superiority; p = 0.907, Proportional Odds Regression; The analysis was not adjusted for baseline factors

6. Secondary Outcome: Rescue Medication Use
Description: Number of participants using rescue medication during the 8-hour follow-up period
Time Frame: 8 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine Alone | Lidocaine + Guanfacine
Number analyzed (Participants) | 36 | 28
Participants
  0 hours | 16 | 12
  0.5 hours: number analyzed (Participants) | 35 | 26
  0.5 hours | 2 | 0
  1 hour: number analyzed (Participants) | 34 | 26
  1 hour | 0 | 1
  1.5 hours: number analyzed (Participants) | 30 | 24
  1.5 hours | 3 | 1
  2 hours: number analyzed (Participants) | 30 | 26
  2 hours | 3 | 0
  2.5 hours: number analyzed (Participants) | 30 | 24
  2.5 hours | 1 | 2
  3 hours: number analyzed (Participants) | 31 | 25
  3 hours | 4 | 3
  3.5 hours: number analyzed (Participants) | 30 | 24
  3.5 hours | 1 | 1
  4 hours: number analyzed (Participants) | 31 | 26
  4 hours | 1 | 1
  4.5 hours: number analyzed (Participants) | 24 | 21
  4.5 hours | 3 | 2
  5 hours: number analyzed (Participants) | 32 | 25
  5 hours | 3 | 2
  5.5 hours: number analyzed (Participants) | 28 | 25
  5.5 hours | 2 | 1
  6 hours: number analyzed (Participants) | 32 | 26
  6 hours | 2 | 1
  6.5 hours: number analyzed (Participants) | 31 | 26
  6.5 hours | 1 | 3
  7 hours: number analyzed (Participants) | 29 | 24
  7 hours | 3 | 2
  7.5 hours: number analyzed (Participants) | 27 | 26
  7.5 hours | 5 | 2
  8 hours | 7 | 1
Statistical Analysis 1: Comparison: Lidocaine Alone vs Lidocaine + Guanfacine; Test type: Superiority; p = 0.373, Regression, Logistic; Adjusted for use of pain medication at baseline

7. Secondary Outcome: Time to First Rescue Medication
Description: Time, in hours, to use of first rescue medication in the follow-up period following the injection.
Time Frame: 14 days
Population: Not all participants reported using rescue medication, so this analysis only includes participants that reported rescue medication use.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Lidocaine Alone | Lidocaine + Guanfacine
Number analyzed (Participants) | 30 | 23
hours | 10.28 (23.54) | 23.76 (60.89)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks after injection
Arm/Group | Lidocaine Alone | Lidocaine + Guanfacine
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/28
Other Adverse Events (participants affected / at risk) | 2/36 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine Alone (N=36) | Lidocaine + Guanfacine (N=28)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Left ear pressure after procedure (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Facial brusing and sensitivity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT03865940/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03865940/ICF_000.pdf